CLINICAL TRIAL: NCT06642675
Title: Effectiveness of Navigated Transcranial Magnetic Stimulation (nTMS) of Left Supramarginal Gyrus for Negative Symptoms : A Double-blind, Randomized Controlled Trial
Brief Title: nTMS for Negative Symptom in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: nTMS
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia; TMS; negative symptom
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group: active iTBS (Experimental): Patients assigned to experimental group would receive treatment of active iTBS. 50 iTBS sessions (1,800 pulses per session, 50-minute intersession interval) were delivered 10 days at 90% resting motor threshold.
  Interventions: Device: Intermittent theta burst stimulation(iTBS)
- control group: sham iTBS (Sham Comparator): Patients assigned to control group would receive treatment of sham iTBS. The iTBS mode in sham iTBS is as the same as the active iTBS, but would be delivered with the sham coil, which provides the sensation of TBS without enough magnetic energy to reach the cortex.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Intermittent theta burst stimulation(iTBS) — By using the TMS Navigation System, the iTBS will be targeted at the left Supramarginal Gyrus.iTBS will be performed using Magstim Rapid² stimulator, parameters are set to triplet 50Hz bursts, repeat at 5Hz, 2s seconds on and 8 seconds off, 1800 pulses per session, intensity of 90% resting motor threshold(RMT), total duration of 10 minutes.
  Other Names: Navigated transcranial magnetic stimulation (nTMS)
  Arms: experimental group: active iTBS
Device: Sham stimulation — Patients in sham group would receive the same intervention procedure as the active ITBS group, but the coil will be replaced with sham coil, which provides the sensation of TBS without enough magnetic energy to reach the cortex.
  Arms: control group: sham iTBS

SUMMARY:
This research aims to test the effectiveness of Navigated transcranial magnetic stimulation (nTMS) of left Supramarginal Gyrus for negative symptoms. In this double-blind, randomized controlled trial, patients will be assigned to active iTBS experimental group or sham iTBS group. Treatment will last for 10 days, and data will be collected at baseline, 1 day and 1 month after treatment.

DETAILED DESCRIPTION:
This research aims to test the effectiveness of Navigated transcranial magnetic stimulation (nTMS) for negative symptoms in patients with schizophrenia. In this double-blind, randomized controlled trial, patients will be assigned to active iTBS experimental group or sham iTBS group. By using the TMS Navigation System, the iTBS will be targeted at the left Supramarginal Gyrus, and parameters are set to triplet 50Hz bursts, repeat at 5Hz, 2s seconds on and 8 seconds off, 1800 pulses per session, intensity of 90% resting motor threshold(RMT), total duration of 10 minutes.Both group will receive nTMS 5 times a day, total treatment for 10 days. Measurements included a pretreatment measurement session, 10 days of nTMS treatment, a post-treatment measurement, and a follow-up measurement 1 month after treatment. At baseline, data of demographic variables (such as sex, age, years of education, occupational status, social support) and disease characteristics (such as duration of illness, antipsychotic daily dose in chlorpromazine equivalents, family psychiatric history) will be collected.At baseline, the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7) , data of outcomes (such as Positive and Negative Symptom Scale (PANSS) score,Negative Symptoms(SANS) score and other secondary outcomes) will be collected in order to test the effectiveness of nTMS. After completing the 1 month follow-up, patients may choose whether to continue follow-up , in order to observe the long-term effects of the treatment. However, they will not receive any further experimental interventions.

ELIGIBILITY:
Inclusion Criteria:

* 1.Clinical diagnosis of schizophrenia according to ICD-11.
* 2.Confirmation of the diagnosis of schizophrenia using the SCID-5-RV (DSM-5 Structured Clinical Interview for DSM-5 Disorders - Research Version).
* 3.Score more than 4 points on either item of negative symptoms (N1-N7).
* 4.Aged less than 60 years.

Exclusion Criteria:

* 1.Clinical diagnosis or SCID-5-RV assessment confirming neurodevelopmental disorders, bipolar and related disorders, substance use disorders (excluding alcohol and tobacco).
* 2.Presence of severe or acute physical illnesses, including traumatic brain injury, intracranial space-occupying or infectious diseases, acute cardiovascular diseases, acute respiratory system diseases, acute hematological disorders, etc.
* 3.Presence of clearly defined genetic diseases, including tuberous sclerosis, multiple sclerosis, Kleefstra syndrome, 22q11.2 deletion syndrome, Prader-Willi syndrome, Klinefelter syndrome (47,XXY), etc.
* 4.Contraindication for MRI examination or rTMS, such as metal implantation in the body, epilepsy, cochlear implants, etc.
* 5.Severe risk of self-injury or suicide
* 6.Other conditions where the researchers find unsuitable for the treatment

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Positive and Negative Symptom Scale (PANSS) score | Baseline, the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7)
  The PANSS measures positive symptoms, negative symptoms and general psychopathology. It contains 30 items, each item is scored from 1 to 7, higher score indicates more severe psychopathology in the dimension. Here the investigators use the Chinese version of the PANSS to evaluate the severity of symptoms in schizophrenia in different participant and different treatment phase. The investigators mainly focus on change in the total score of the negative symptoms.
Change in Scale for Assessment of Negative Symptoms(SANS) score | Baseline, the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7)
  The SANS measures the severity of negative symptoms in schizophrenia. It contains 24 items, each item is scored from 0 to 5, higher score indicates more severe symptom. The SANS evaluates five dimensions of the negative symptoms, which are apathy, poverty of thought, abulia, social withdrawal and disorders of attention.

SECONDARY OUTCOMES:
Change in MATRICS Consensus Cognitive Battery (MCCB) score | Baseline, the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7)
  The MCCB measures the cognitive function in schizophrenia and other neuropsychiatric diseases. It covers nine cognitive domains including attention, information processing speed, verbal learning and memory, visual learning and memory, spatial working memory, reasoning, problem solving, social cognition, executive function and fine motor. Raw scores are converted to scale scores, then to normalized T scores. T scores of seven domains and composite score are further calculated. The changes of scores at different follow up timepoint will be used for assessing the improvement of cognitive function (higher score means a better outcome).
The data of head resting-state functional magnetic resonance imaging | Baseline, the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7)
  All patients undergo head MRI scans in Siemens Trio 3.0T scanner. Resting functional MRI will be acquired based on Blood Oxygenation Level Dependent (BOLD) contrast. It can detect changes in blood oxygenation to analyze the change of brain function after intervention.
Change in Personal and Social Performance Scale (PSP) score | Baseline, the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7)
  The PSP is a 100-point single-item rating scale that assesses four important domains of patients with mental disorders : (a) socially useful activities, including work and study, (b) personal and social relationships, (c) self-care, and (d) disturbing and aggressive behaviors. Higher score indicates better social function.
Change in Global Assessment Function (GAF) score | Baseline, the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7)
  The GAF is a 100-point single-item rating scale that evaluate level of patients with schizophrenia, combining the level of social function and the severity of psychiatric symptoms to produce a single score. Higher score indicates better social function.
Change of electroencephalogram | Baseline, first day of treatment (day 1), the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7)
  Neuroscan multi-channel evoked potential workstation records EEG data, using the international 10-20 system for electrode placement, with Ag/AgCl electrodes on a 64/128 electrode cap.
Change of TMS-EEG (Transcranial Magnetic Stimulation Electroencephal | Baseline, the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7)
  Neuroscan multi-channel evoked potential workstation records EEG data, using the international 10-20 system for electrode placement, with Ag/AgCl electrodes on a 64/128 electrode cap. During TMS-EEG recording, stimulation of 100 single TMS pulses were delivered at 100% RMT intensity while participants remained at rest with their eyes open.
Change in Montgomery-Asberg Depression Rating Scale (MADRS) score | Baseline, the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7)
  MADRS is a 10-item scale that measures the severity of depression symptoms. Each item is scored from 0 to 6, higher score indicates more severe symptom.
Change in Calgary Depression Scale for Schizophrenia (CDSS) score | Baseline, the day of the end of treatment (day 11±1), 1 month after the treatment (day40±7)
  CDSS is a nine item clinician rated outcome measure that assesses the level of depression in people with schizophrenia. Each item is scored from 0 to 3, higher score indicates more severe symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, M.D., Ph.D., Study Chair — Mental Health Institute of Second Xiangya Hospital,CSU
Locations (1):
- Mental Health Institute of Second Xiangya Hospital,CSU, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No